CLINICAL TRIAL: NCT03627702
Title: The Effect of VIP Light on Healing Bedsores Process
Brief Title: Treatment of Bedsores With VIP Light
Status: Completed | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Jolanta Zwolińska, Assistant professor, University of Rzeszow
Other Study IDs: Piler
Record Dates: First submitted 2018-05-26; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Light; Therapy; Bedsore
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All bedsores were irradiated with a Bioptron lamp. Photo and measurement of bedsores size and Torrance score, were made: on the first, 9,18 and 36 day of therapy.
  Interventions: Radiation: Irradiated VIP (Visible Incoherent Polarized)

INTERVENTIONS:
Radiation: Irradiated VIP (Visible Incoherent Polarized) — 20 irradiations were performed twice a day. The exposure time was 10 minutes. Exposure was made at a distance of 10 cm.

SUMMARY:
Difficulty healing wounds have a significant effect to the general fitness of the patient and his quality of life. On Account of the frequency of their appearing, constitute the serious health and social problem. In comprehensive dealing with such patients physiotherapy will matter greatly. The visible polychromatic polarized light is most often used physical factor assisting comprehensive treatment bedsores.

Purpose of the work: Analyze of using the visible polychromatic polarized light in the comprehensive process of healing bedsores at elderly people with the limited motor activity.

Material and methods: Participants receive interventions as part of routine medical care, and a researcher studies the effect of the intervention. The study was conducted in people over 65 years old, with bedsores grade III and IV in Torrance scale. The therapy included radiation of bedsores with VIP light. Effectiveness of the method of treatment was examined using photographic images and to measure the extent of the wound.

DETAILED DESCRIPTION:
18 people were examined. In all subjects, were assessed the risk of developing bedsores according to the scale Dutch Consensus Prevention of Bedsores CBO. All bedsores were irradiated with a Bioptron lamp (20 sessions, twice a day). Photo and measurement of bedsores size and Torrance score, were made:on the first, 9, 18 and 36 day of therapy.

ELIGIBILITY:
Inclusion Criteria:

* a high risk of bedsores development (Dutch Consensus Prevention of Bedsores CBO)
* having a bedsore(s)
* permanent stay in a nursing home
* recommended light therapy (VIP light)

Exclusion Criteria:

* ability to locomotion
* age under 65 years old

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
scale Dutch Consensus Prevention of Bedsores CBO | The first day of the therapy (one measure)
  Scale Dutch Consensus Prevention of Bedsores CBO - score on a scale of 0 to 3 points of mental state, neurological status, ability to move, nutritional status, way of eating, function of the anal sphincters and urethra, age, body temperature, medicines, comorbid diabetes. 8 points or more indicate a risk of bedsores.
Bedsores classification: the Torrance system | Change is being assessed after 36 days
  Assessment of the degree damage and color of tissue.
  1°-the lowest degree of bedsore 5°- the highest degree of bedsore
Measurement of bedsores size | Change is being assessed after 36 days
  Vertical and horizontal size of bedsores

SECONDARY OUTCOMES:
Photo of bedsores | On the first, 9, 18 and 36 day of therapy
  Visual image of bedsores

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Zwolińska, PhD, Principal Investigator — University of Rzeszow

IPD SHARING:
Plan to Share IPD: No
Lack of consent of participants due to difficult contact

REFERENCES:
- [Background] Bhattacharya S, Mishra RK. Pressure ulcers: Current understanding and newer modalities of treatment. Indian J Plast Surg. 2015 Jan-Apr;48(1):4-16. doi: 10.4103/0970-0358.155260. PMID 25991879
- [Result] Thomas E, Vinodkumar S, Mathew S, Setia MS. A Study of the Factors Associated with Risk for Development of Pressure Ulcers: A Longitudinal Analysis. Indian J Dermatol. 2015 Nov-Dec;60(6):566-72. doi: 10.4103/0019-5154.169127. PMID 26677269
- [Result] Rutteman B, Borremans K, Beckers J, Devleeschouwer E, Lampmann S, Corthouts I, Verlinde P. Aeromonas wound infection in a healthy boy, and wound healing with polarized light. JMM Case Rep. 2017 Oct 16;4(10):e005118. doi: 10.1099/jmmcr.0.005118. eCollection 2017 Oct. PMID 29188066
- [Result] Oliveira PC, Pinheiro AL, de Castro IC, Reis JA Jr, Noia MP, Gurgel C, Teixeira Cangussu MC, Pedreira Ramalho LM. Evaluation of the effects of polarized light (lambda400-200 nm) on the healing of third-degree burns in induced diabetic and nondiabetic rats. Photomed Laser Surg. 2011 Sep;29(9):619-25. doi: 10.1089/pho.2010.2914. Epub 2011 Jun 1. PMID 21631376
- [Result] Pinheiro AL, Meireles GC, Carvalho CM, de Barros Vieira AL, dos Santos JN, Ramalho LM. Biomodulative effects of polarized light on the healing of cutaneous wounds on nourished and undernourished Wistar rats. Photomed Laser Surg. 2006 Oct;24(5):616-24. doi: 10.1089/pho.2006.24.616. PMID 17069493
- [Result] Ishmamet'ev II, Deriabin EI, Zharov VV, Ishmamet'ev IL, Tochilova ER. [Microcirculation changes after polarized polychromatic light use in preoperative period in cases of face cosmetic operations]. Stomatologiia (Mosk). 2008;87(6):38-40. Russian. PMID 19156105
- [Result] Akilbekova D, Boddupalli A, Bratlie KM. The effect of polarized light on the organization of collagen secreted by fibroblasts. Lasers Med Sci. 2018 Apr;33(3):539-547. doi: 10.1007/s10103-017-2398-0. Epub 2017 Nov 30. PMID 29192340
- [Result] Tada K, Ikeda K, Tomita K. Effect of polarized light emitting diode irradiation on wound healing. J Trauma. 2009 Nov;67(5):1073-9. doi: 10.1097/TA.0b013e318187ad02. PMID 19680158
- See also: Pressure ulcers - physiotherapy in the treatment process — http://evereth.pl/odlezyny-fizjoterapia-w-procesie-leczenia/